CLINICAL TRIAL: NCT07196397
Title: POL-CA Registry: Multicenter Observational Study of Neuromodulatory Procedures in Cardiovascular Autonomic Dysfunction Syndromes
Brief Title: POLish Registry of CArdioneuroablation and CArdioneuromodulation
Acronym: POL-CA
Status: Recruiting | Type: Observational
Sponsor: SABAMED Medical Center Ltd. (Network)
Responsible Party: Sponsor
Other Study IDs: 51/2024/В
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Vasovagal Syndrome VVS; Cardioinhibitory Carotid Sinus Syndrome CSS; Symptomatic Sinus Bradycardia SB or Atrioventricular Block AV; Postural Orthostatic Tachycardia Syndrome POTS; Orthostatic Hypotension; Inappropriate Sinus Tachycardia Syndrome IST; Vasospastic Angina; Microvascular Angina; Ventricular Arrythmia; Raynaud Phenomena; Autonomic Dysfunction; Autonomic Diseases
Keywords: cardioneuroablation; cardiac sympathetic denervation; sinoatrial node sparing hybrid ablation; catheter ablation; neural stimulation; cardioneuromodulation; percutaneus stellate ganglion blockage; cardiac rehabilitation; cardiovascular autonomic tests; syncope
MeSH Terms: conditions — Hypotension, Orthostatic; Angina Pectoris, Variant; Microvascular Angina; Primary Dysautonomias; Autonomic Nervous System Diseases; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- vagally mediated bradycardia: This cohort includes patients with vagally mediated bradycardia, including cardioinhibitory vasovagal syncope, carotid sinus syndrome, or functional sinus node dysfunction related to excessive parasympathetic activation. Patients are referred for interventional treatment due to recurrent syncope or symptomatic bradycardia refractory to conservative management. Interventions include cardioneuroablation or autonomic modulation procedures aimed at reducing vagal influence on the sinus and atrioventricular nodes while preserving physiological autonomic balance. Diagnosis is confirmed based on tilt-table testing, ECG documentation, and symptom correlation.
  Interventions: Procedure: cardioneuroablation; Behavioral: Hybrid Cardiac Rehabilitation Program
- IST/POTS: This cohort includes patients diagnosed with inappropriate sinus tachycardia (IST) or postural orthostatic tachycardia syndrome (POTS) who are undergoing interventional treatment due to insufficient response to pharmacological or behavioral therapy. Interventions include sinus node-sparing thoracoscopic ablation aimed at improving symptoms and quality of life. Autonomic dysfunction is confirmed based on standardized testing, and the interventions target neural pathways involved in excessive sympathetic or inadequate parasympathetic control of heart rate and vascular tone.
  Interventions: Procedure: SN sparing hybrid ablation; Behavioral: Hybrid Cardiac Rehabilitation Program; Device: Transcutaneous Vagus Nerve Stimulation (tVNS)
- Cardiac sympathetic denervation: Patients with clinical indications for stand-alone or concomittant, hybrid cardiac sympathetic denervation. This cohort includes patients with arrhythmias driven by excessive sympathetic activation, such as congenital long QT syndrome (LQTS), catecholaminergic polymorphic ventricular tachycardia (CPVT), and refractory ventricular tachyarrhythmias. Patients are referred for cardiac sympathetic denervation (CSD) due to high arrhythmic burden despite optimal pharmacologic treatment or recurrent implantable cardioverter-defibrillator (ICD) shocks. CSD is performed via thoracoscopic access and involves ablation or removal of the stellate ganglion and thoracic sympathetic chain (typically T2-T4). The goal is to reduce sympathetic drive, stabilize cardiac electrophysiology, and prevent life-threatening arrhythmias.
  Interventions: Procedure: Cardiac sympathetic denervation; Behavioral: Hybrid Cardiac Rehabilitation Program
- other rare subgroups and neuromodulation intervention: This cohort includes patients with rare autonomic or electrophysiological syndromes undergoing neuromodulatory interventions as part of individualized treatment strategies. Interventions may include transcutaneous vagus nerve stimulation (tVNS), structured cardiac rehabilitation programs with autonomic modulation components, and other non-invasive or minimally invasive techniques aimed at improving autonomic balance and symptom burden. This group is characterized by heterogeneous diagnoses, including overlapping or atypical forms of autonomic dysfunction, and is managed with a personalized, multidisciplinary approach integrating physiologic monitoring, rehabilitation, and neuromodulation.
  Interventions: Procedure: cardioneuroablation; Procedure: SN sparing hybrid ablation; Procedure: Cardiac sympathetic denervation; Behavioral: Hybrid Cardiac Rehabilitation Program; Device: Transcutaneous Vagus Nerve Stimulation (tVNS)

INTERVENTIONS:
Procedure: cardioneuroablation — Cardioneuroablation and related autonomic interventions aim to modulate parasympathetic and/or sympathetic inputs to the heart in order to treat functional bradycardia, inappropriate sinus tachycardia, vasovagal syncope, and other reflex arrhythmias. Techniques include catheter-based ablation of ganglionated plexi, thoracoscopic sinus node-sparing ablation, cardiac sympathetic denervation, and percutaneous stellate ganglion blockade. These procedures are tailored to each patient's autonomic profile and diagnosis.
  Groups: other rare subgroups and neuromodulation intervention; vagally mediated bradycardia
Procedure: SN sparing hybrid ablation — Sinus node-sparing hybrid ablation is a minimally invasive surgical procedure that modulates autonomic inputs to the sinoatrial node while preserving its intrinsic function. The intervention is performed via video-assisted thoracoscopic surgery (VATS) and targets the epicardial autonomic ganglia and neural connections responsible for inappropriate sinus tachycardia or autonomic dysfunction. Unlike traditional sinus node modification, this approach avoids direct ablation of the sinus node and focuses on surrounding autonomic structures. The goal is to reduce pathologic chronotropic activity and improve symptom control without inducing iatrogenic bradycardia.
  Groups: IST/POTS; other rare subgroups and neuromodulation intervention
Procedure: Cardiac sympathetic denervation — Cardiac sympathetic denervation is an interventional procedure aimed at reducing excessive sympathetic drive to the heart by ablating or removing components of the sympathetic nervous system. It is typically performed via a thoracoscopic approach and involves bilateral or left-sided denervation of the stellate ganglion and thoracic sympathetic chain (usually T2-T4). CSD is used in patients with arrhythmias associated with sympathetic overactivity, such as long QT syndrome, catecholaminergic polymorphic ventricular tachycardia (CPVT), or autonomic dysfunction-related tachyarrhythmias. The procedure helps reduce arrhythmic burden, modulate autonomic tone, and improve symptom control.
  Groups: Cardiac sympathetic denervation; other rare subgroups and neuromodulation intervention
Behavioral: Hybrid Cardiac Rehabilitation Program — A two-phase program combining supervised inpatient exercise, respiratory training, psychological support, and education with a home-based telerehabilitation phase (Nordic walking, remote ECG and vital sign monitoring). The aim is to restore functional capacity, reduce symptoms, and improve autonomic balance.
Device: Transcutaneous Vagus Nerve Stimulation (tVNS) — Transcutaneous vagus nerve stimulation (tVNS) is a non-invasive neuromodulation technique in which the vagus nerve is stimulated via surface electrodes placed on the skin, most commonly in the auricular region (e.g., tragus or cymba conchae). The intervention is performed using a certified external stimulation device that delivers mild electrical impulses to activate afferent vagal fibers. tVNS is used in the treatment of various conditions, including depression, epilepsy, migraine, chronic pain, and disorders of the autonomic nervous system such as postural orthostatic tachycardia syndrome (POTS) and inappropriate sinus tachycardia (IST). In this study, tVNS is applied as a supportive neuromodulatory therapy with individualized stimulation parameters and session duration based on clinical response and patient tolerance.
  Groups: IST/POTS; other rare subgroups and neuromodulation intervention

SUMMARY:
The multicentre observational study POL-CA involves a wide spectrum of patients with a history of syncopy. The study recruits patients with diagnosed vasovagal syndrome, cardioinhibitory carotid sinus syndrome, symptomatic sinus bradycardia or atrioventricular block, postural orthostatic tachycardia syndrome, orthostatic hypotension, and inappropriate sinus tachycardia syndrome. This is an observational, controlled study with retrospective, clinical data analysis of previously treated patients and the analysis of syncopal patients prospectively recruited into the study. The aim of the POL-CA registry is to create a platform for physicians to record treatment data for patients undergoing procedures that affect innervation or modify cardiovascular reflexes (cardioneuroablation, cardioneuromodulation) in order to provide a multicentre summary of population characteristics and treatment outcomes based on a standardized POL-CA questionnaire and methodology for various arrhythmias.

DETAILED DESCRIPTION:
The study aims to include a group of at least 1,000 individuals, taking into account subgroups of patients with rare diseases involving fewer than 50 individuals (e.g., carotid sinus hypersensitivity or familial sinus bradycardia). Participants will be divided into three age groups: 18-40 years, 41-60 years, and over 60 years. These individuals will undergo procedures affecting innervation or modifying cardiovascular reflexes (cardioneuroablation or neuromodulation) due to ineffective pharmacological treatment or training methods. This group will also include patients who, according to guidelines, qualify for pacemaker implantation but declined the procedure.

The clinical trial protocol specifies inclusion and exclusion criteria. The protocol outlines the collection of various data, including traditional medical history (including contact information) and data related to the interventional treatment performed (including assessment of treatment efficacy and the occurrence of both perioperative and long-term complications). Additionally, the protocol includes the use of scales and questionnaires to evaluate patient symptoms and well-being, as well as an analysis of standard and non-standard verbal and non-verbal behaviors of patients. Scales and questionnaires used to assess patient symptoms and well-being: EQ-5D, SF-36, VASIS for bradycardia symptoms (daytime, before sleep, nighttime, and morning), and MALMO scoring test.

Patients will also routinely undergo physical performance evaluations (assessment using the Borg scale, HRR analysis, correlation of heart rate values during exercise before and after the procedure, 6MWT walk tests, and analysis of tele-rehabilitation outcomes).

Patient follow-up will be conducted at 1, 6, and 12 months post-procedure and then annually from 2024 to 2030, with ECG evaluations. The primary endpoint of the study is the spontaneous recurrence of symptoms that were present before the procedure affecting innervation and/or cardiovascular reflexes.

Enrolment in the POL-CA registry does not involve performing any additional invasive medical procedures on the patients.

The Single POL-CA Registry for a specific treatment technique will be managed by an appointed project leader. The project leader will be responsible for preparing a literature review, inclusion criteria, and clinical and electrophysiological characteristics of the given treatment technique. The project leader either becomes the first author of the publication or designates one. Physicians' participation in the project will be voluntary, with acceptance of audits or data verification at local centres. Patient personal data will only be accessible to the local investigator and will remain protected. The order of authorship for the publication will be determined based on the contributions of the other project participants (e.g., number of patients, manuscript preparation, data analysis).

The POL-CA online platform will include a standardized data creation panel for the project leader and the study's website. Data collection will comply with standard encryption, protection procedures, and the requirements of bioethics and scientific committees.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of at least one of the following conditions:

  * Inappropriate sinus tachycardia (IST)
  * Postural orthostatic tachycardia syndrome (POTS)
  * Vasovagal syncope (VVS)
  * Cardioinhibitory carotid sinus syndrome (CSS)
  * Symptomatic sinus bradycardia or functional AV block
  * Orthostatic hypotension (OH)
* History of recurrent autonomic symptoms (e.g., syncope, bradycardia, palpitations, orthostatic intolerance)
* Undergoing or previously underwent interventional treatment affecting cardiac autonomic innervation (e.g., cardioneuroablation, SN-sparing ablation, cardiac sympathetic denervation)
* Provided written informed consent (for prospective arm)

Exclusion Criteria:

* Structural heart disease requiring surgical intervention
* Permanent pacemaker or ICD implanted prior to enrollment
* Inability to complete follow-up assessments or questionnaires
* Severe psychiatric comorbidities impairing participation
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years and older with documented autonomic cardiovascular dysfunction, referred for or previously treated with procedures targeting cardiac innervation. The population includes both men and women, and covers a broad clinical spectrum including IST, POTS, VVS, CSS, sinus bradycardia, and orthostatic hypotension. Participants are enrolled across multiple centers in Poland. The study includes both retrospective and prospective cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Recurrence of Pre-Treatment Autonomic Symptoms at 12 Months | Baseline and 1, 6, and 12 months post-intervention
  Recurrence is defined as the spontaneous return of autonomic symptoms (e.g., syncope, orthostatic intolerance, palpitations, bradycardia) that were present before the intervention. Symptoms are confirmed by clinical assessment, structured questionnaires (e.g., VASIS, MALMO, EQ-5D), and ECG data. This outcome will help evaluate the long-term effectiveness of autonomic modulation procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Stec, Prof., MD, PhD, Principal Investigator — SABAMED Medical Center Ltd.; Marta Kornaszewska, MD, Study Director — SABAMED Medical Center Ltd.
Locations (1):
- SabaMed, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the registry collects sensitive clinical information on rare cardiovascular autonomic disorders. Only aggregated, de-identified summary results will be reported in scientific publications and presentations. Access to raw patient-level data will remain restricted to local investigators in compliance with GDPR and bioethics committee requirements.

REFERENCES:
- [Background] Ahmed A, Charate R, Bawa D, Ghazal R, Garg J, Pothineni NVK, Kabra R, Della Rocca DG, Atkins D, Lakkireddy P, Bommana S, Al-Ahmad A, Shenthar J, Padmanabhan D, Narasimhan C, DiBiase L, Romeya A, Gopinathannair R, Natale A, Lakkireddy D. Bilateral Cardiac Sympathetic Denervation for Refractory Multifocal Premature Ventricular Contractions in Patients With Nonischemic Cardiomyopathy. JACC Clin Electrophysiol. 2024 Jan;10(1):31-39. doi: 10.1016/j.jacep.2023.09.014. Epub 2023 Nov 8. PMID 37943190
- [Background] Stec S, Kuteszko R, Sulik A, Kornaszewska M. Double trouble: Hybrid management of inappropriate sinus tachycardia and sinus bradycardia in the era of cardioneuromodulation. HeartRhythm Case Rep. 2025 Aug 16;11(11):1151-1156. doi: 10.1016/j.hrcr.2025.08.012. eCollection 2025 Nov. No abstract available. PMID 41333861
- [Background] Kornaszewska M, Wilczek-Banc A, Ratajska A, Piotrowicz E, Szkaradek B, Kowalewski M, Suwalski P, Ogorzelec N, Wileczek A, Zajac M, Pastyrzak M, Stec S. Implementation of a Hybrid Cardiac Rehabilitation and Symptom Scoring System in Patients with Inappropriate or Postural Sinus Tachycardia Referred for Sinus Node Sparing Hybrid Ablation. J Clin Med. 2025 Aug 20;14(16):5879. doi: 10.3390/jcm14165879. PMID 40869705
- [Background] Stec S, Suwalski P, de Asmundis C, La Meir M, Reichert A, Wilczek-Banc A, Szkaradek B, Kowalewski M. EP-Heart Team approach with sinus node sparing ablation for complex inappropriate sinus tachycardia and postural orthostatic tachycardia syndrome: A first experience in Central Europe. Kardiol Pol. 2025;83(3):342-344. doi: 10.33963/v.phj.103819. Epub 2025 Jan 2. No abstract available. PMID 39743902
- [Background] de Asmundis C, Pannone L, Lakkireddy D, Beaver TM, Brodt CR, Lee RJ, Frazier K, Chierchia GB, La Meir M. Hybrid epicardial and endocardial sinus node-sparing ablation therapy for inappropriate sinus tachycardia: Rationale and design of the multicenter HEAL-IST IDE trial. Heart Rhythm O2. 2023 Jan 31;4(4):275-282. doi: 10.1016/j.hroo.2023.01.005. eCollection 2023 Apr. PMID 37124558
- [Background] Lakkireddy D, Garg J, DeAsmundis C, LaMeier M, Romeya A, Vanmeetren J, Park P, Tummala R, Koerber S, Vasamreddy C, Shah A, Shivamurthy P, Frazier K, Awasthi Y, Chierchia GB, Atkins D, Bommana S, Di Biase L, Al-Ahmad A, Natale A, Gopinathannair R. Sinus Node Sparing Hybrid Thoracoscopic Ablation Outcomes in Patients with Inappropriate Sinus Tachycardia (SUSRUTA-IST) Registry. Heart Rhythm. 2022 Jan;19(1):30-38. doi: 10.1016/j.hrthm.2021.07.010. Epub 2021 Jul 30. PMID 34339847
- [Background] Aksu T, Brignole M, Calo L, Debruyne P, Di Biase L, Deharo JC, Fanciulli A, Fedorowski A, Kulakowski P, Morillo C, Moya A, Piotrowski R, Stec S, Sutton R, van Dijk JG, Wichterle D, Tse HF, Yao Y, Sheldon RS, Vaseghi M, Pachon JC, Scanavacca M, Meyer C, Amin R, Gupta D, Magnano M, Malik V, Schauerte P, Shen WK, Acosta JCZ. Cardioneuroablation for the treatment of reflex syncope and functional bradyarrhythmias: A Scientific Statement of the European Heart Rhythm Association (EHRA) of the ESC, the Heart Rhythm Society (HRS), the Asia Pacific Heart Rhythm Society (APHRS) and the Latin American Heart Rhythm Society (LAHRS). Europace. 2024 Aug 3;26(8):euae206. doi: 10.1093/europace/euae206. PMID 39082698
- [Background] Kulakowski P, Baran J, Sikorska A, Krynski T, Niedzwiedz M, Soszynska M, Piotrowski R. Cardioneuroablation for reflex asystolic syncope: Mid-term safety, efficacy, and patient's acceptance. Heart Rhythm. 2024 Mar;21(3):282-291. doi: 10.1016/j.hrthm.2023.11.022. Epub 2023 Nov 29. PMID 38036236
- [Background] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133
- [Background] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Background] Tomasiewicz K, Woron J, Kobayashi A, Krasinski Z, Rydzewska G, Szymanski FM. Post-COVID-19 syndrome in everyday clinical practice: interdisciplinary expert position statement endorsed by the Polish Society of Civilization Diseases. Pol Arch Intern Med. 2024 May 28;134(5):16728. doi: 10.20452/pamw.16728. Epub 2024 Apr 15. PMID 38619233
- [Background] Spahic JM, Hamrefors V, Johansson M, Ricci F, Melander O, Sutton R, Fedorowski A. Malmo POTS symptom score: Assessing symptom burden in postural orthostatic tachycardia syndrome. J Intern Med. 2023 Jan;293(1):91-99. doi: 10.1111/joim.13566. Epub 2022 Sep 16. PMID 36111700
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Aug 20;74(7):e51-e156. doi: 10.1016/j.jacc.2018.10.044. Epub 2018 Nov 6. No abstract available. PMID 30412709
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. Practical Instructions for the 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):e43-e80. doi: 10.1093/eurheartj/ehy071. No abstract available. PMID 29562291
- [Background] Ajijola OA, Aksu T, Arora R, Biaggioni I, Chen PS, De Ferrari G, Dusi V, Fudim M, Goldberger JJ, Green AL, Herring N, Khalsa SS, Kumar R, Lakatta E, Mehra R, Meyer C, Po S, Stavrakis S, Somers VK, Tan AY, Valderrabano M, Shivkumar K. Clinical neurocardiology: defining the value of neuroscience-based cardiovascular therapeutics - 2024 update. J Physiol. 2025 Mar;603(7):1781-1839. doi: 10.1113/JP284741. Epub 2025 Mar 8. PMID 40056025